CLINICAL TRIAL: NCT07230665
Title: Outcome of Patients With Malignant Gastric Outlet Obstruction Undergoing Endoscopic Ultrasound-guided Gastroenterostomy or Enteral Metal Stenting: a Prospective Cohort Study
Brief Title: Outcome of Patients With Malignant Gastric Outlet Obstruction Undergoing Endoscopic Ultrasound-guided Gastroenterostomy or Enteral Metal Stenting
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Principal Investigator, National Taiwan University Hospital
Other Study IDs: 202108046RINC
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Gastric Outlet Obstruction Due to Malignancy; EUS Guided Enteroenteric Anastomosis; Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic enteral stent placement: This procedure was performed under fluoroscopic guidance. Either a duodenoscope or a forward-viewing therapeutic endoscope was used to access the obstruction. A 0.025-or 0.035-inch guidewire was advanced into the jejunum beyond the obstruction using a 20mm extraction balloon catheter. After positioning the catheter across the stricture, contrast was injected to determine the location and length of the stricture. An uncovered, through-the-scope duodenal stent (BONASTENT; Standard Sci Tech, Seoul, Korea or WallFlex; Boston Scientific, Marlborough, Mass, USA) with a diameter of 22 mm and a length of 6 to 16 cm, depending on the stricture length, was then deployed to adequately cover both ends of the obstruction under combined fluoroscopic and endoscopic guidance.
  Interventions: Procedure: Endoscopic ultrasound-guided gastroenterostomy

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided gastroenterostomy — This procedure was performed under general anesthesia with endotracheal intubation. After identifying the site and extent of the obstruction similar with ES, a 7Fr nasobiliary drain was advanced over the guidewire into the target jejunum under fluoroscopic guidance. A linear echoendoscope was then advanced into the stomach to visualize the jejunum. The jejunal loop was adequately distended by continuously infusing a mixture of saline, contrast medium, and indigo carmine using a standard water pump. Once the target jejunum was confirmed, an antispasmodic was administered. Using the freehand technique, the gastric and jejunal walls were directly punctured with an electrocautery- enhanced LAMS (Hot AXIOS, 20 mm diameter, 10 mm length; Boston Scientific). The LAMS was deployed under EUS and fluoroscopic guidance-first the distal flange into the jejunum, followed by intrachannel release of the proximal flange within the echoendoscope, and then its advancement outside the working channel.

SUMMARY:
Gastric outlet obstruction (GOO) refers to a mechanical blockage of the distal stomach or duodenum that prevents normal passage of food and liquids. According to literature, 50-80% of GOO cases are caused by malignant tumors compressing or directly invading the gastrointestinal tract. Among patients with pancreatic cancer, 15-20% develop GOO [1,2]. GOO is also considered a poor prognostic factor in malignancy, with a median survival time of only 3-6 months [3].

Traditionally, management options for GOO include surgical gastrojejunostomy and endoscopic enteral metal stent (ES) placement. Endoscopic approaches are less invasive, allow earlier oral intake, and reduce hospital stay [4-6]. Considering that most patients with malignant GOO are debilitated, a less invasive option is often preferable.

In recent years, endoscopic ultrasound-guided gastroenterostomy (EUS-GE) has emerged as an alternative. A recent systematic review and meta-analysis comparing ES and EUS-GE found similar technical and clinical success rates, but significantly lower re-intervention rates in the EUS-GE group [7]. However, most existing studies are retrospective and lack systematic, prospective follow-up data comparing the two approaches remain lacking.

This study aims to prospectively evaluate and compare the short- and long-term outcomes-including stent function, oral intake, nutritional status, and quality of life-of patients with malignant GOO undergoing either EUS-GE or conventional enteral stenting.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 18 years or older who underwent ES or EUS-GE for unresectable mGOO were enrolled

Exclusion Criteria:

* Prior enteral stent placement
* Multi-level bowel obstruction,
* Linitis plastica of the stomach
* A life expectancy of less than one mont
* Uncorrected coagulopathy
* Pregnancy
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter prospective study involved 13 academic centers in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reintervention rate | one year
  Defined as the need for additional endoscopic treatment due to recurrent GOO symptoms

SECONDARY OUTCOMES:
Technical success | one year
  Successful stent placement across or bypass the obstruction, confirmed by endoscopy or fluoroscopy
Clinical success | one year
  1. ≥ 2 point improvement in the gastric outlet obstruction score (GOOS) after stent insertion;
  2. GOOS categorized oral intake into four levels (the minimum and maximum score from 0 to 3): 0 (fasting), 1 (liquid diet), 2 (soft diet), and 3 (normal/low-residue diet).
Gastric outlet obstruction score (GOOS) changes | one year
  1. GOOS categorized oral intake into four levels (the minimum and maximum score from 0 to 3): 0 (fasting), 1 (liquid diet), 2 (soft diet), and 3 (normal/low-residue diet).
  2. Comparison the GOOS change before and after stent placement (GOOS recored while the patients was discharge)
Adverse events (AEs) | one year
  AEs, including stent misdeployement, perforation, and bleeding, were classified and graded according to the Adverse Events in GI Endoscopy (AGREE) classification, with a 30-day cut-off distinguishing early and late events.
Survival | one year
  alive until the last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Nataional Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided